CLINICAL TRIAL: NCT07315802
Title: A Prospective Study on a New Pattern of Retinal Laser Treatment for Proliferative Diabetic Retinopathy (PDR)
Brief Title: New Pattern of Retinal Laser Treatment for PDR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Retinal Laser for PDR
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Proliferative Diabetic Retinopathy; Photocoagulation Burn to Retina

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Retinal laser (Experimental): This is a single arm study using literature-reported outcomes of PDR patients as the comparator.
  Interventions: Procedure: A new pattern of retinal laser

INTERVENTIONS:
Procedure: A new pattern of retinal laser — A new pattern of retinal argon laser combines anti VEGF treatment within 2 weeks. Spot argon-laser photocoagulation was started 1 disc-diameter nasal to the optic disc, outside the superior and inferior vascular arcades, and 2 disc diameter (DD) temporal to the fovea, and the mid-peripheral retina flanking the large vessels. Further peripheral PRP and anti-VEGF administration would be added only if neovascularization progress.

SUMMARY:
The objective of the study is to evaluate the efficacy of a new pattern of argon-laser in treating patients with proliferative diabetic retinopathy (PDR).

DETAILED DESCRIPTION:
Argon-laser pan retinal photocoagulation (PRP) is the first-line therapy for proliferative diabetic retinopathy (PDR) nowadays, which is believed to function by reducing retinal ischemia and decreasing the stimulation for neovascularization. However, diabetic retinopathy (DR) would still progress uncontrollably even after PRP, and PRP would result in reduction in visual acuity and loss of peripheral visual field, which may be influenced by the distribution pattern of the retinal laser treatment.

A variety of modified argon-laser patterns have been reported - a more central PRP, a more peripheral PRP, a central-sparing PRP or an extended-targeted PRP, yet the risk of developing neovascularization is higher in retina around the posterior vascular arcades and alongside the major retinal vessels.

This study will include 300 patients with PDR, who will be treated with a new pattern of argon-laser. An initial retinal laser would be given in the posterior retina outside the arcades and the mid-peripheral retina flanking the large vessels. Then investigators will conduct no less than 2 years follow-up. Further peripheral PRP and anti-VEGF administration would be added only if neovascularization progress, aiming to stop DR progression with the minimum of laser energy.

ELIGIBILITY:
Inclusion Criteria:

1. Having given free and informed consent to take part in the study.
2. Diabetes mellitus (DM) under stable treatment during the study, aged 18y to 70y, with no significant underlying systemic diseases (such as impaired renal function, severe cardiac disease, etc.);
3. Clinically diagnosed PDR, with the presence of neovascularization confirmed by ultra-widefield fundus photography and widefield OCT angiography.

Exclusion Criteria:

1. Previous treatment with PRP;
2. Previous treatment with anti-VEGF agents or corticosteroids within 3 months;

2. Severe cataract, massive vitreous hemorrhage, or extensive preretinal hemorrhage that makes pan retinal photocoagulation impossible; 3. Unable to tolerate argon-laser retinal treatment.; 4. Vitreous macular traction or traction retinal detachment need to be performed with vitrectomy; 5. Retinal vascular occlusion, age-related macular degeneration, retinal angioma, uveitis, glaucoma, optic neuropathy, or other ocular diseases that can lead to vitreous hemorrhage and/or neovascularization; 6. Other conditions that the researcher found improper to be included into this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
BCVA | From enrollment to the end of the 2-year follow-up period. (at enrollment; 1 month, 3months, 6 months, 1 year and 2 years after the initial laser treatment)
  BCVA stands for best-corrected visual acuity, measured by Snellen chart.
CMT | From enrollment to the end of the 2-year follow-up period. (at enrollment; 1 month, 3months, 6 months, 1 year and 2 years after the initial laser treatment)
  CMT stands for central macular thickness, measured with optical coherence tomography (OCT) images, which serves as one of the key indicators of DR progression.
Mean VF loss | 1 year and 2 years after the initial laser treatment during the follow-up period.
  VF stands for visual field. Mean deviation would be used to evaluate the VF loss.
Further treatment | From enrollment to the end of the 2-year follow-up period.
  Number of participants with further laser treatment, anti-VEGF treatment or vitrectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye and ENT Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided